CLINICAL TRIAL: NCT02417922
Title: The Effect of Autologous Conditioned Plasma Treatment for Conservative Treated Total Achilles Tendon Tears: Randomized Double Blinded Placebo Control Trial
Brief Title: Effect of Autologous Conditioned Plasma Treatment for Conservative Treated Total Achilles Tendon Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anders Ploug Boesen, Medical Doctor, Bispebjerg Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1-2010-052
Record Dates: First submitted 2011-12-08; First posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Tendon Rupture
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous conditioned plasma (ACP) (Experimental): Whole blood was drawn from the patients using arthrex system (total of 10 mls whole blood). After that whole blood spinning is conducted for 5 minutes and ACP with platelets and growth factors is separated from the red and white blood cells (around 4 mls).
  ACP is injected at baseline, 2 weeks, 4 weeks and after 6 weeks from injury date.
  Interventions: Other: ACP
- Saline (Placebo Comparator): Saline (4 mls) is injected around the ruptured achilles tendon at baseline, 2 weeks, 4 weeks and after 6 weeks from injury date.
  Interventions: Other: Saline

INTERVENTIONS:
Other: Saline — 4 mls of saline is injected 4 times around the injured tendon area every 2nd week during the 8 weeks of conservative treatment.
  Arms: Saline
Other: ACP — 4 mls of ACP is injected 4 times around the injured tendon area every 2nd week during the 8 weeks of conservative treatment.
  Arms: Autologous conditioned plasma (ACP)

SUMMARY:
The purpose is to see if Autologous Conditioned Plasma (ACP) promote and accelerating tendon tissue healing in Conservative treated total Achilles Tendon Tears.

40 healthy males were randomized to either receive ACP or Placebo (saline) around the ruptured achilles tendon at baseline, 2 weeks, 4 weeks and again after 6 weeks during the 8 weeks immobilization period with an orthosis. Ultrasound and symptoms scores (ATLS) was performed at baseline, after 8 weeks immobilization and again after 3 month, 6 month and 12 month. Scoring and functional tests was performed after the 8 weeks immobilization and again after 12 weeks, 24 weeks and 52 weeks from injury date.

DETAILED DESCRIPTION:
Total achilles rupture is a severe injury and many has long lasting functional deficit afterwards. Treatment options is either operative or conservative treatment. Conservative treatment for total Achilles rupture has become more and more popular during the last 10 years. Nevertheless we still see a higher risk of re-rupture compared to surgery.

Aim: The aim of the study is in patients with acute total Achilles tendon rupture to examine if Autologous Conditioned Plasma (ACP) promote and accelerate tendon tissue healing in Conservative treated total Achilles tendon rupture and thereby gives a better functional outcome.

Materials and methods: Healthy males (25-60 years; n=40) with acute total achilles tendon ruptures is randomly assigned to either 1) ACP (~ 4 mls) or 2) placebo (saline ~ 4 mls) treatment. Participants will be treated on 4 successive occasions with 2 weeks (wks) interval during the 8 week conservative treatment with an orthoses. The injections will be performed under ultrasound guidance. All subjects will undergo a 8 weeks immobilization period with an orthoses with full weigh bearing and after that they will be guided in a proper rehabilitation regime during the intervention. Clinical effects will be assessed as changes in functional scoring system (ATLS), isometric muscle strength and muscle function (one-legged heel-rise test). Furthermore tendon length will be measured by ultrasound. All outcome measures will be recorded at baseline and again after 8 weeks immobilization (expect muscle strength and function), 12 weeks, 24 weeks and 52 weeks after injury.

Results: Look at possible changes and differences between groups (ACP and Placebo) in ATLS scores, muscle strength, ultrasound tendon length elongation and muscle function.

Statistics: All data will be analyzed in SigmaPlot v11 using two-way repeated measures ANOVA with Student-Newman-Keuls Post-hoc test. This is used to see changes over time in all groups (time effect) and differences between groups within time-points (group effect). All data will be presented as mean ± SEM time.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-60 years.
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.
* The patient should be able to follow the instructed regimen with a removable ankle orthosis.
* The patient must be able to determine when rupture occurred, and it can't be over 4 days old.
* The patient should be able to follow the postoperative controls.

Exclusion Criteria:

* Terminal illness.
* Former achilles tendon rupture
* Former surgery on the achilles tendon
* Treatment with fluoroquinolones during the last 6 months.
* Tendinosis treated with a tablet or injection with corticosteroids within the last 6 months.
* Diagnosis of arterial insufficient in the leg.
* Lack of palpable pulse in the foot
* Severe medical illness: ASA score greater than 2

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
ATRS (Achilles Tendon Total Rupture Score) | After immobilization period (8 weeks) and again after 12 weeks, 24 weeks and 52 weeks from injury date
  Patient-reported validated scoring tool developed for assessment of symptoms and physical activity after treatment for acute achilles tendon rupture (score 0-100 points)

SECONDARY OUTCOMES:
Isometric Strength test | After 12 weeks, 24 weeks and 52 weeks from injury date
  The subjects were asked to produce an isometric contraction of the calf muscle with increasing force to their maximum voluntary effort (MVC) over a 10 sec period. The MVC was performed on both legs to measure the differences between the two legs.
Heel-rise test | After 12 weeks, 24 weeks and 52 weeks from injury date
  The accumulated work made doing repetitive heel-rises is measured on each leg to see the differences between the two legs.
Tendon elongation | At baseline, after immobilization (8 weeks) and again after 12 weeks, 24 weeks and 52 weeks from injury date
  Tendon length was measured with ultrasound on both legs during intervention to see possible tendon elongation after achilles rupture. The landmarks for measure the tendon length was the proximal part of the top of the calcaneus bone and most distal part of the muscular-tendinous part of the m. gastrocnemius medial.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, Dr. Med., Principal Investigator — Institute of Sportsmedicine Copenhagen, Bispebjerg Hospital
Locations (1):
- Institute of Sportsmedicine, Bispebjerg hospital, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Boesen AP, Boesen MI, Hansen R, Barfod KW, Lenskjold A, Malliaras P, Langberg H. Effect of Platelet-Rich Plasma on Nonsurgically Treated Acute Achilles Tendon Ruptures: A Randomized, Double-Blinded Prospective Study. Am J Sports Med. 2020 Jul;48(9):2268-2276. doi: 10.1177/0363546520922541. Epub 2020 Jun 2. PMID 32485112